CLINICAL TRIAL: NCT00349388
Title: A Randomized Trial Comparing Once Daily Dosing vs. Multiple Doses a Day of Mesalamine in Pediatric Patients With Quiescent Ulcerative Colitis
Brief Title: Safety and Compliance of Taking Mesalamine Once a Day in Pediatric Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: none enrolled in second arm, therfore no analysis
Sponsor: Annette Langseder (Other)
Collaborators: Procter and Gamble (Industry)
Responsible Party: Sponsor-Investigator, Annette Langseder, Joel Rosh, MD, Atlantic Health System
Organization: Atlantic Health System (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R05-11-010
Record Dates: First submitted 2006-07-05; First posted 2006-07-07 (Estimated); Results first posted 2014-08-15 (Estimated); Last update posted 2019-01-29 (Actual); Status verified 2019-01

CONDITIONS: Ulcerative Colitis
Keywords: Mesalamine; Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Mesalamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Asacol once a day dosing (Experimental): Asacol total dose in mg/kg given once a day
  Interventions: Drug: Asacol
- Asacol BID/TID dosing (Active Comparator): Asacol total dose split BID or TID
  Interventions: Drug: Asacol

INTERVENTIONS:
Drug: Asacol — Asacol is given once a day versus twice or three times a day
  Other Names: Mesallamine

SUMMARY:
To determine whether once a day administration of Mesalamine is at least as safe and efficacious and administration of multiple doses a day in preventing clinical relapse of ulcerative colitis in children and adolescence.

DETAILED DESCRIPTION:
Is taking total dose in mg/kg once a day, as safe as taking total dose divided in mg/kg spreadout during the day in preventing clinical relapse of ulcerative colitis in children and adolescence.

ELIGIBILITY:
Inclusion Criteria:

* Ages 6 to 18 years,
* Must be able to swallow tablets, and
* Biopsy proven ulcerative colitis

Exclusion Criteria:

* Allergy or hypersensitivity to Mesalamine or other salicylates
* Use of rectal medications

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1 (Actual)
Dates: Start 2006-07; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joel Rosh, MD, Principal Investigator — Atlantic Health System
Locations (1):
- Morristown Memorial Hospital/Goyerb Children's Hospital, Morristown, New Jersey, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Asacol Once a Day Dosing | Asacol BID/TID Dosing
Started | 0 (no patients enrolled) | 1
Completed | 0 (no patients enrolled , therefore no patients completed) | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: No patients enrolled into intervention arm due to lack of enrollment.Only 1 subject was enrolled in Control arm. Therefore no data can be compared for study outcome
Groups:
- Total: Total of all reporting groups
Arm/Group | Asacol Once a Day Dosing | Asacol BID/TID Dosing | Total
Number analyzed (Participants) | 0 | 1 | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years |  | 1 | 1
  Between 18 and 65 years |  | 0 | 0
  >=65 years |  | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female |  | 0 | 0
  Male |  | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States |  | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Once Daily Dosing Works as Well a Multiple Dosing a Day.
Description: subject tolerated once a day dose Only 1 subject enrolled which was the control arm standard dose twice a day. No subjects enrolled to take dose once a day Therefore, primary outcome cannot be reported
Time Frame: overall study
Population: cannot analysze primary outcome because no subjects were enrolled in the once a day dose arm. Study was terminated due to lack of enrollment
Arm/Group | Asacol Once a Day Dosing | Asacol BID/TID Dosing
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Improved Medication Compliance.
Description: Not applicable : unable to measure secondary outcome because no one was enrolled in once a day dose arm. Therefore, no comparisons can be made to see if once a day dosing would have higher compliance than taking medication BID or TID
Time Frame: overall study
Population: Not applicable: unable to measure secondary outcome because no one was enrolled in once a day dose arm. Therefore, no comparisons can be made to see if once a day dosing would have a higher compliance than taking medication BID or TID. Study was terminated due to lack of enrollment.
Measure: Count of Participants; unit: Participants
Arm/Group | Asacol Once a Day Dosing | Asacol BID/TID Dosing
Number analyzed (Participants) | 0 | 1
Participants | 0 | 1

ADVERSE EVENTS:
Time Frame: 180 days total
Description: No subjects were enrolled in the once daily dosing arm. Therefore, no subject was at risk for Serious Adverse Events or non Serious Events
Arm/Group | Asacol Once a Day Dosing | Asacol BID/TID Dosing
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/1
Other Adverse Events (participants affected / at risk) | 0/0 | 0/1

LIMITATIONS AND CAVEATS:
No subjects were analysed due to lack of enrollment. No subject was enrolled into the once a day dosing arm to answer our primary or secondary outcomes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes